CLINICAL TRIAL: NCT05848921
Title: Research on Changes of Cerebral Vascular Morphology and Cognitive Function in Patients With Carotid Artery Stenosis Before and After Surgery
Brief Title: Evaluation of Brain Health and Surgical Efficacy in Patients With Carotid Artery Stenosis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Nanjing University of Traditional Chinese Medicine (Other)
Collaborators: Xi'an Jiaotong University (Other); The 2rd School of Medicine，WMU/The 2rd Affiliated Hospital and Yuying Children's Hospiyal of WMU (Unknown)
Responsible Party: Principal Investigator, Qianyan Liu, Principal Investgator, Nanjing University of Traditional Chinese Medicine
Other Study IDs: 82071993-2
Record Dates: First submitted 2023-04-28; First posted 2023-05-08 (Actual); Last update posted 2023-05-08 (Actual); Status verified 2023-04

CONDITIONS: Carotid Artery Stenosis; Image
Keywords: Carotid Artery Stenosis; MRI Imaging
MeSH Terms: conditions — Carotid Stenosis | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- CAS-CN: Carotid Artery Stenosis with cognitive normality
  Interventions: Device: magnetic resonance image; Diagnostic Test: Neuropsychological scale
- CAS-MCI: Carotid Artery Stenosis with mild cognitive impairment
  Interventions: Device: magnetic resonance image; Diagnostic Test: Neuropsychological scale
- HC: Healthy controls
  Interventions: Device: magnetic resonance image; Diagnostic Test: Neuropsychological scale

INTERVENTIONS:
Device: magnetic resonance image — Imaging data were collected in a strong magnetic field
Diagnostic Test: Neuropsychological scale — Multi dimensional neuropsychological test

SUMMARY:
The purpose of this study is to explore the relationship between the recovery of cerebrovascular morphology and cognitive function before and after surgical treatment in patients with carotid artery stenosis and their preoperative cardiac health status. And combined with preoperative cognitive status, serum markers, and cardiovascular health evaluation indicators, evaluate and predict the possibility of postoperative neurodegenerative diseases and the level of cerebrovascular health in patients.

DETAILED DESCRIPTION:
The aim of this study is to evaluate the brain health status and surgical efficacy of patients with carotid artery stenosis. Firstly, investigate whether hemodynamic parameters such as blood flow reserve fraction at the carotid artery stenosis site are correlated with white matter hyperintensities and cerebral vascular morphological changes in elderly patients with normal cognition and mild cognitive impairment; Then, when the blood flow of carotid artery has been improved after surgery, compare the cerebrovascular health of patients before surgery and the way of cerebral vascular reconstruction; Combined with the postoperative neuropsychological cognitive test to explore the postoperative cognitive recovery of patients, and combined with the postoperative imaging data and the biomarker in the blood of patients at various stages, to explore the way of cerebral vascular reconstruction and changes in brain structure and function of different groups of patients behind cognitive changes.

ELIGIBILITY:
Inclusion Criteria:

* Aged over 50 years old;
* Conscious and capable of completing neuropsychological scales
* Clinical detection of carotid artery stenosis requires surgical treatment;
* Compliant with carotid artery stenting or carotid endarterectomy surgical standards
* Individuals with normal cognition and mild cognitive impairment

Exclusion Criteria:

* Degree of vascular blockage in other intracranial segments ≥ 50%
* Have a history of mental illness, nervous system disease (such as stroke) or brain injury with loss of consciousness for more than five minutes;
* Neurological and psychiatric disorders unrelated to AD (schizophrenia, depression, etc.), post-traumatic stress disorder, obsessive-compulsive disorder, multiple sclerosis, amyotrophic lateral sclerosis)
* Have a history of alcohol or drug abuse
* There are contraindications for magnetic resonance imaging examination
* Those with significant organ dysfunction such as lung, liver, and kidney;
* Patients with intracranial tumors, infectious diseases, and blood system diseases;
* Participating in other clinical studies at the same time

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All of the patients of carotid artery stenosis group are in-patients and out-patients in the cardiac surgery department from the research center. The subjects of control group are recruited from community.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-05-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change of brain volume before and after treatment | before operation; 3-10 Days after operation; 1 month; 6-12months]
  The change of brain volume (mm3) are evaluated by structural 3DT1 weighted MRI. Freesurfer software is used to get the measured value of the volume.
Change of cerebrovascular morphology before and after treatment | before operation; 3-10 Days after operation; 1 month; 6-12months
  The change of Cerebral vessel density, caliber and tortuosity, brain white matter hyperintensity lesion count
Change of brain function connectivity before and after operation | before operation; 3-10 Days after operation; 1 month; 6-12months
  The change of brain functional connectivity intensity are evaluated by rest stage functional MRI. DPABI software based on MATLAB is used to get the measured the matrix value of functional connectivity.

SECONDARY OUTCOMES:
Change of serum marker concentration before and after operation | before operation; 3-10 Days after operation; 1 month; 6-12months
  The change of serum marker concentration is evaluated by inflammatory cytokine.
Change of plasma marker concentration before and after operation | before operation; 3-10 Days after operation; 1 month; 6-12months
  The change of plasma marker concentration is evaluated by neurofilament light chain(NFL) protein extracted from plasma.
Brain evaluate basic cognition before operation | before operation
  Basic cognition is evaluated by Mini-mental State Examination (MMSE) and Clinical Dementia Rating (CDR) . For MMSE , The minimum value is 0 , and the maximum value is 30. The higher scores mean a better outcome. For CDR , the results are represented by scores of 0,0.5,1,2,3, and the degree of cognitive impairment is classified as normal, suspicious, mild, moderate, and severe
Change of executive functions before and after operation evaluated by Trail-Making Test Part A | before operation; 3-10 Days after operation; 1 month; 6-12months
  The change of executive functions are first evaluated by Trail-Making Test Part A test. The minimum value is 0 , and the maximum value is 30. This test has no clear maximum and minimum values. If the test completion time exceeds 79 seconds, it means the outcome is abnormal. The higher scores mean a worse outcome.
Change of executive functions before and after operation evaluated by Digit Symbol Coding score | before operation; 3-10 Days after operation; 1 month; 6-12months
  The change of executive functions are second evaluated by Digit Symbol Coding score. The minimum value is 0 , and the maximum value is not clear. The normal range of results is 56.53 ± 20.17. The higher scores mean a better outcome.
Change of working memory before and after operation evaluated by Forward Digit Span | before operation; 3-10 Days after operation; 1 month; 6-12months
  The change of working memory is first evaluated by Forward Digit Span. The minimum value is 0 , and the maximum value is not clear. The normal range of results is 7.75±1.47. The higher scores mean a better outcome.
Change of working memory before and after operation evaluated by Backward Digit Span | before operation; 3-10 Days after operation; 1 month; 6-12months
  The change of working memory is second evaluated by Backward Digit Span. The minimum value is 0 , and the maximum value is not clear. The normal range of results is 5.36±1.91. The higher scores mean a better outcome.
Change of language function before and after operation evaluated by Language Fluency test | before operation; 3-10 Days after operation; 1 month; 6-12months
  The change of language function is evaluated by Language Fluency test. The minimum value is 0 , and the maximum value is not clear. The normal range of results is 19.43±4.81. The higher scores mean a better outcome.
Change of executive functions before and after operation evaluated by Clock Drawing Test | before operation; 3-10 Days after operation; 1 month; 6-12months
  The change of executive functions is evaluated by Backward Digit Span. The minimum value is 0 , the maximum value is 4.
Change of executive functions before and after operation evaluated by Trail-Making Test Part B | before operation; 3-10 Days after operation; 1 month; 6-12months
  The change of executive functions are first evaluated by Trail-Making Test Part B test. The minimum value is 0 , and the maximum value is 30. This test has no clear maximum and minimum values. If the test completion time exceeds 79 seconds, it means the outcome is abnormal. The higher scores mean a worse outcome.It is a supplement to Trail-Making Test Part A, which is optional for patients who are not familiar with the English alphabetical order

CONTACTS AND LOCATIONS:
Overall Officials: Bo Yin, phD, Principal Investigator — The 2rd School of Medicine，WMU/The 2rd Affiliated Hospital and Yuying Children's Hospiyal of WMU
Locations (1):
- The 2rd School of Medicine，WMU/The 2rd Affiliated Hospital and Yuying Children's Hospiyal of WMU, Wenzhou, Zhejiang, China